CLINICAL TRIAL: NCT07267546
Title: Heart-Lung Machine: Impact of the Priming Solution on the Body's Acid-Base Balance, Electrolyte Composition and Clinical Outcome (PRIMEII)
Brief Title: Heart-Lung Machine: Impact of the Priming Solution on Acid-Base Balance, Electrolytes and Outcome on Patients Undergoing Cardiac Surgery
Acronym: PRIMEII
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2025-02925-01-749040
Record Dates: First submitted 2025-11-17; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Acid Base Imbalance; Osmolality Disturbance; Crystalloid Solutions; Electrolyte Changes; Cardiopulmonary Bypass
Keywords: cardiopulmonary bypass; priming solution; acid base balance; electrolytes; plasma osmolality
MeSH Terms: conditions — Acid-Base Imbalance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Ringer's Acetate 80 (Active Comparator): Ringer's Acetate 1100 ml with addition of 80 mmol NaCl
  Interventions: Diagnostic Test: Ringer's Acetate 80
- Plasmalyte (Active Comparator): Plasmalyte 1100 ml, no addition
  Interventions: Diagnostic Test: Plasmalyte
- Ringer's Acetate no add (Active Comparator): Ringer's Acetate 1100 ml, no addition
  Interventions: Diagnostic Test: Ringer's Acetate no add
- Ringer's Acetate 160 (Active Comparator): Ringer's Acetate with addition of 160 mmol NaCl
  Interventions: Diagnostic Test: Ringer's Acetate 160

INTERVENTIONS:
Diagnostic Test: Ringer's Acetate 80 — Cardiopulmonary bypass circuit will be primed with Ringer's Acetate 1100 ml and 80 mmol NaCl
  Arms: Ringer's Acetate 80
Diagnostic Test: Plasmalyte — Cardiopulmonary bypass circuit will be primed with Plasmalyte 1100 ml, no addition.
  Arms: Plasmalyte
Diagnostic Test: Ringer's Acetate no add — Cardiopulmonary bypass circuit will be primed with Ringer's Acetate 1100 ml no addition
  Arms: Ringer's Acetate no add
Diagnostic Test: Ringer's Acetate 160 — Cardiopulmonary bypass circuit will be primed with Ringer's Acetate 1100 ml and 160 mmol NaCl
  Arms: Ringer's Acetate 160

SUMMARY:
Most cardiac surgery procedures requires the use of heart-lung machine. The heart-lung machine circuit needs to be filled with a fluid before connecting it to the patients circulation. This is called priming and is accomplished by filling the circuit with a solution used for fluid replacement. The circuit in our institution requires 1100 mL to be filled.

The body has several mechanisms with the purpose to maintain its state of balance. When a large amount of clear solution suddenly enters the blood stream this balance can be altered. The goal of this clinical trial is to investigate different priming solutions in the heart-lung machine circuit. The main questions it aims to answer are:

How do different priming solutions alter the acid-base balance, osmolality and electrolytes which reflects the body's water balance for patients undergoing cardiac surgery with the use of heart-lung machine?

There will be 4 different groups:

1. Ringer-Acetate, 1100 mL / no addition
2. Ringer-Acetate, 1100 mL + 80 mmol sodium chloride (NaCl)
3. Ringer-Acetate, 1100 mL + 160 mmol NaCl
4. Plasmalyte, 1100 mL / no addition Blood samples will be taken before, during and after surgery, post operative day 1 and 4 to analyze acid-base balance, electrolytes, and plasma osmolality. Urine output and hydration status will also be collected until post operative day 1. After 3 months, a blood sample will be taken for analysis of electrolytes and kidney function.

DETAILED DESCRIPTION:
Cardiopulmonary bypass (CBP) with a heart-lung machine is mandatory for a vast majority of cardiac surgeries. Briefly the disposables in a CPB circuit consists of a reservoir, an oxygenator and tubings.

The role of CPB can be summarized as follows:

1. Empty the heart. Drain out the blood (achieved via venous cannulas).
2. Oxygenate the blood and remove carbon dioxide. Thus, the lungs are not participating during CPB.
3. Maintain homeostasis and adjust chemical and electrolyte blood composition.
4. Maintain or adjust the body's temperature via a heat exchanger, which is a part of the heart-lung machine.
5. Return oxygenated blood to the patient via arterial cannula.

Heart-lung machine provides even the following:

1. Salvage blood loss during surgery via cardiotomy suckers and return it to the patient.
2. Prevent distention of the heart during surgery via cardiac vents.
3. Deliver cardioplegia which stops the heart, providing myocardial protection and condition to perform cardiac surgery.
4. Additional treatments, such as hemofiltration and removing av cytokines.

Before connecting the CPB circuit to the patient's circulation it needs to be deaired. This is achieved by priming, i.e. filling the circuit with a liquid solution. The 2024 EACTS (European Association for Cardio-Thoracic Surgery)/EACTA (European Association of Cardiothoracic Anaesthesiology)/EBCP (European Board of Cardiovascular Perfusin) Guidelines on CPB in adult cardiac surgery point out that despite a wealth of studies, no consensus has been reached on the optimal composition of the priming solution. According to recent surveys, balanced crystalloids are the preferred priming solution, but there are no recommendations of the composition in the solution. The standard prime solution at our institution consists of Ringer Acetate which is a common crystalloid fluid in Sweden used intravenously for fluid and volume loss. Due to its composition, i.e. lower pH and sodium and higher chloride concentrations than the human blood, it is sometimes necessary to add electrolytes and other components to the circuit either in advance or after initiation of CPB. Previous studies have investigated various prime compositions and plasma osmolality. The crystalloid priming fluid used in these studies contained mannitol, which has a high osmolality. A former study from our group showed a significant decrease in blood sodium with a mannitol-containing prime, but no effects on plasma osmolality. Highly osmolar priming solution has further been studied, also containing mannitol, and found a steep rise in plasma osmolality. These studies used priming fluids with an addition of 80 mmol NaCl and 160 mmol NaCl, respectively. Plasmalyte is a newer crystalloid solution with a composition of sodium and chloride more similar to human plasma which could be of advantage. Plasmalyte is used for CPB priming in some cardiac centers. Studies on Plasmalyte as a priming solution have shown less metabolic acidosis compared to Ringer Lactate. However, it has not been used in our institution for this purpose and there are no studies comparing Plasmalyte with Ringer Acetate. The literature search has further not found any studies investigating non-mannitol CPB priming solutions with differing additions of NaCl. There is a need to fill this knowledge gap to proceed in developing of the optimal priming solution, tailored to variouse preexisting diseases or conditions.

Scientific questions The overall aim of the project is to investigate if clinical outcome after cardiac surgery can be improved by optimizing the priming solution.

The sub-projects will answer the questions:

* Do the different priming solutions: Ringer Acetate alone, Ringer Acetate with added NaCl and Plasmalyte alone affect the acid-base balance and composition of electrolytes in the blood?
* Do the different priming solutions affect the need to correct the acid-base balance during the heart-lung machine period?
* Do the different priming solutions affect the total fluid balance in connection with cardiac surgery?
* Do the different priming solutions affect the osmolality in the blood per- and postoperatively?
* Do the different priming solutions affect postoperative renal function? Do the different priming solutions affect neurological outcome?

ELIGIBILITY:
Inclusion Criteria:

* Patients 18 years and above
* Undergoing coronary artery bypass graft (CABG) surgery as single surgery
* Undergoing aortic valve replacement (AVR) as single surgery (AtriClip is allowed)
* Given consent to participate, both verbal and written

Exclusion Criteria:

* Subnormal heart function (defined as an ejection fraction <45%), and no signs of heart failure (edema).
* Body weight <60 kg or >120 kg
* Preoperative hemoglobin <120 g/L,
* Subnormal kidney function (defined as GFR <30 ml/min),
* Blood sodium outside normal range (135-145 mmol/l),
* Need of acute surgery
* AVR due to aortic valve insufficiency
* Changes in operating method or addition of intraoperative procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Acid Base Balance | Measurements will be taken at anesthesia induction, 3 minutes after administration of cardioplegia, 30 minutes after onset of CPB, 5 minutes after termination of CPB, 1 hour post operative, day 1 and day 4 post operative.
  This study uses blood samples that are taken at predefined timepoints
Sodium concentration | Measurements will be taken at anesthesia induction, 3 minutes after administration of cardioplegia, 30 minutes after onset of CPB, 5 minutes after termination of CPB, 1 hour post operative, day 1 and day 4 post operative, and at month 3.
  This study uses blood samples that are taken at predefined timepoints
Osmolality | Measurements will be taken at anesthesia induction, 3 minutes after administration of cardioplegia, 30 minutes after onset of CPB, 15 minutes after termination of CPB, 1 hour post operative, day 1 and day 4 post operative
  This study uses blood samples that are taken at predefined timepoints

SECONDARY OUTCOMES:
Chloride, magnesium -and potassium concentrations | Measurements will be taken at anesthesia induction, 3 minutes after administration of cardioplegia, 30 minutes after onset of CPB, 5 minutes after termination of CPB, 1 hour post operative, day 1 and day 4 post operative, and at month 3.
  This study uses blood samples that are taken at predefined timepoints
Urine output | Measurements of urine output will be registered during cardiac surgery and 24 hours post operative.
  Production of urine will be studied during cardiac operation and post operative
Kidney function | Blood samples will be collected pre operative - the day before surgery or in morning the same day, 1 hour post operative, day 1 and day 4 post operative, and at month 3.
  Creatinine-and urea concentration, glomerular filtration rate
Neurological outcome | Blood samples will be collected at anesthesia induction, 1 hour post operative, day 1 and day 4 post operative.
  S-100, a prognostic biomarker used for assessing brain injury

CONTACTS AND LOCATIONS:
Overall Officials: Snejana Hyllén, Phd,MD, Principal Investigator — Region Skane
Locations (1):
- Skane University hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Anonymized participant data can be made available on request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Anonymized data will be available November 2026 and stored for 10 years.
Access Criteria: Requests must be from studies with appropriate ethics approval.

REFERENCES:
- [Background] Surabhi S, Kumar M. Comparison of ringer's lactate and plasmalyt-a as cardiopulmonary bypass prime for bypass associated acidosis in valve replacement surgeries. Ann Card Anaesth. 2021 Jan-Mar;24(1):36-41. doi: 10.4103/aca.ACA_104_19. PMID 33938829
- [Background] Ljunggren M, Skold A, Dardashti A, Hyllen S. The use of mannitol in cardiopulmonary bypass prime solution-Prospective randomized double-blind clinical trial. Acta Anaesthesiol Scand. 2019 Nov;63(10):1298-1305. doi: 10.1111/aas.13445. Epub 2019 Jul 29. PMID 31287556
- [Background] Malmqvist G, Claesson Lingehall H, Appelblad M, Svenmarker S. Cardiopulmonary bypass prime composition: beyond crystalloids versus colloids. Perfusion. 2019 Mar;34(2):130-135. doi: 10.1177/0267659118793249. Epub 2018 Aug 16. PMID 30114960
- [Background] Wahba A, Kunst G, De Somer F, Agerup Kildahl H, Milne B, Kjellberg G, Bauer A, Beyersdorf F, Berg Ravn H, Debeuckelaere G, Erdoes G, Haumann RG, Gudbjartsson T, Merkle F, Pacini D, Paternoster G, Onorati F, Ranucci M, Ristic N, Vives M, Milojevic M; EACTS/EACTAIC/EBCP Scientific Document Group. 2024 EACTS/EACTAIC/EBCP Guidelines on cardiopulmonary bypass in adult cardiac surgery. Eur J Cardiothorac Surg. 2025 Feb 4;67(2):ezae354. doi: 10.1093/ejcts/ezae354. No abstract available. PMID 39949326